CLINICAL TRIAL: NCT06693583
Title: VR as a Distraction Technique for Management of Acute Anxiety and Pain During Outpatient Colposcopy Procedures - a Single Centre Randomised Control Trial
Brief Title: Mind Over Cervix: Using Virtual Reality to Reduce Colposcopy Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Gateshead Health NHS Foundation Trust (Other); Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FCNUR-23-098
Record Dates: First submitted 2024-02-02; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Anxiety; Colposcopy
Keywords: Colposcopy; Anxiety Reduction; Cervical screening; Virtual Reality; Pain reduction
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Masking Description: Participants will be blindly randomly allocation to the control or intervention arm, however due to the nature of the study it will not be possible to blind the participant or assessor.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm : Standard colposcopy care (No Intervention): Women in the control arm will be offered all aspects of standard colposcopy care for their pain relief. This includes : nursing support, local anaesthetic and gas and air as required.
- Virtual reality headsets as a distraction method (Experimental): The patient will attend for colposcopy at which the consultation will begin as normal. When the time comes for examination +/- biopsy +/- treatment, the patient will be offered the virtual reality headset as a form of immersive therapy to distract them during the procedure. This will be continued until cessation of examination. All other standard forms of pain relief will also be provided for the patient.
  Interventions: Device: Virtual Reality Headsets

INTERVENTIONS:
Device: Virtual Reality Headsets — Virtual reality (VR) headsets are used as a form of distraction technique widely throughout healthcare. Women will be assisted to apply the VR prior to their colposcopy examination beginning. They will be shown an immersive video of walking through a forest that reminds them to breath deeply. The aim is that this will relax them during the colposcopy examination.
  Arms: Virtual reality headsets as a distraction method

SUMMARY:
Colposcopy is an extremely important part of womens healthcare in the prevention of cervical cancer. Women report feeling extremely anxious attending colposcopy, due to the association with cancer and the intimate nature of the examination.

The goal of this clinical trial is to investigate where the use of virtual reality headsets during outpatient colposcopy appointments has any effect on womens' experience. The main question[s] it aims to answer are:

* Does the use of virtual reality headsets reduce anxiety in patients attending colposcopy
* Does the use of virtual reality headsets reduce pain in patients attending colposcopy

Patients will offered to enroll in the trial when they attend for their colposcopy appointment.

Participants will fill out a questionnaire to measure their anxiety beforehand and collect patient demographics.

They will be randomly allocated into the intervention arm or the control arm. This means they will either use virtual reality headset in addition to the standard care, or have standard colposcopy care only After their colposcopy, they will then be asked to to fill out another questionnaire to measure anxiety and pain levels.

If there is a comparison group: Researchers will compare the results from the women who had colposcopy while using the virtual reality headsets to women to see if there is any meaningful difference in anxiety while using the virtual reality headsets.

ELIGIBILITY:
Inclusion Criteria:

* Patients
* women over 18 years of age who attend for outpatient colposcopy and provide informed written consent
* Staff
* Have completed colposcopy training and be a registered member of the British Society of Colposcopy and Cervical Pathology (BSCCP)
* Informed written consent to take part in the trial.

Exclusion Criteria:

* Patients :
* Significant hearing or visual impairments that may effect communication
* Any known characteristics that may make the office procedure more difficult (eg. previous LLETZ, previous cervical conisation, uterine didelphis)
* Inability to provide consent.
* Denial or withdrawal of informed consent orally

Staff :

* The denial or withdrawal of informed consent.
* Trainee colposcopist performing clinic.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Anyone with a cervix who attends for colposcopy.
Enrollment: 141 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
Anxiety level | Before colposcopy and within 15 minutes after the procedure
  Modified State Trait Anxiety Index scores (STAI) will be assessed both prior to colposcopy and afterwards.
  STAI scores is a validated questionaire for measurement of anxiety. It consists of 5 questions with participants self reporting scores. Questions include "I feel frightened," "I feel jittery," " I feel upset," "I feel nervous" and "I feel confused." Outcomes include "Not at all," "Somewhat," "Moderately so" and "very much so." These are scored 1 -4.
  Total scores will range from 5 to 20, with high scores indicating a higher state of anxiety.

SECONDARY OUTCOMES:
Pain level | Within 15 minutes following the procedure
  A numerical rating score from 0-10 will be assess following the procedure for both maximum pain felt and average pain felt.
  Participants will be asked following the colposcopy to rate both the "maximum pain felt, if even for a second," and "average pain felt." This will be measured using a validated Likert scale from 0-10 with 0 indicated no pain, and 10 indicating the worst pain ever felt.

CONTACTS AND LOCATIONS:
Overall Officials: Claire McFeeters, BSc PHd, Study Chair — Universtiy of Ulster
Locations (1):
- Queen Elizabeth Hospital, Gateshead, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All data will be anonymised so no patient identifiable factors will be included in any publications.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT06693583/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-29): https://cdn.clinicaltrials.gov/large-docs/83/NCT06693583/ICF_001.pdf